CLINICAL TRIAL: NCT04463979
Title: Perioperative Evaluation of Cerebellar Tumors: Impact of Cerebellar Functional Topography on Cognition and Motor Ataxia
Brief Title: Perioperative Evaluation of Cerebellar Tumors
Status: Active, not recruiting | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00105872
Record Dates: First submitted 2020-07-02; First posted 2020-07-09 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Cerebellar Tumors; Brain Tumor
MeSH Terms: conditions — Cerebellar Neoplasms; Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cerebellar Tumors: Thirty-three adult (≥18 years of age) patients with primary cerebellar tumors or metastatic tumors located in the cerebellum who will undergo surgery for tumor resection.
  Interventions: Other: Impact of Cerebellar Functional Topography on Cognition and Motor Ataxia
- Brain Tumors: Thirty-three adult (≥18 years of age) patients with primary non-cerebellar brain tumors or metastatic tumors located in a non-cerebellar brain location who will also undergo surgery for tumor resection. This group will be included for comparison.
  Interventions: Other: Impact of Cerebellar Functional Topography on Cognition and Motor Ataxia

INTERVENTIONS:
Other: Impact of Cerebellar Functional Topography on Cognition and Motor Ataxia — Participants in this study will undergo surgical resection of their cerebellar or brain tumor (as per standard of care), as well as clinical and radiographic assessment, including: neurological physical examination (including Karnofsky Performance Scale (KPS) if conducted per Standard of Care), and magnetic resonance imaging (MRI) with or without diffusion tensor imaging (DTI)/tractography, prior to, immediately after, at one-month, 6-month, and 1-year follow-up status post-surgical resection. These data will also be collected at 18-month (±60 days) and 24-month (±60 days) visits post-surgery, if regular office visits with the neurosurgeon are scheduled at these two time points.
  Only at baseline, the following will be conducted: Brief Ataxia Rating Scale (BARS) assessment score, Cerebellar Cognitive Affective Scale (CCAS/Schmahmann syndrome) scale score, Montreal Cognitive Assessment (MoCA) assessment, and a quality of life (QoL) assessment using the SF-36 questionnaire.

SUMMARY:
This is a prospective, cohort study to evaluate the impact of cerebellar functional topography on perioperative outcomes related to cognition and motor ataxia in patients with cerebellar tumors.

DETAILED DESCRIPTION:
Purpose of the Study: This is a prospective, cohort study to evaluate the impact of cerebellar functional topography on perioperative outcomes related to cognition and motor ataxia in patients with cerebellar tumors.

Primary Aim: The primary aim of this study is to determine if patients with a cerebellar tumor are more likely to test positive for cerebellar cognitive affective syndrome than patients with non-cerebellar tumors. This information will be used to improve perioperative assessment in patients with tumors of the cerebellum.

Secondary Aim: To determine the impact of tumor location and cerebellar functional topography on perioperative outcomes (determined by standard of care neurological evaluation and brain images) in patients undergoing resection of cerebellar tumors. This information will be used to improve perioperative assessment in patients with tumors of the cerebellum.

Study Interventions: Thirty-three adult (≥18 years of age) patients with primary cerebellar brain tumors or metastatic brain tumors located in the cerebellum who will undergo surgery for tumor resection, and 33 adult patients with primary non-cerebellar brain tumors or metastatic tumors located in a non-cerebellar brain location who will also undergo surgery for tumor resection will be included in this study. The non-cerebellar brain tumor control group will be included for comparison. Participants in this study will undergo surgical resection of their cerebellar or brain tumor (as per standard of care), as well as clinical and radiographic assessment, including: neurological physical examination (including Karnofsky Performance Scale (KPS) if conducted per Standard of Care), and magnetic resonance imaging (MRI) with or without diffusion tensor imaging (DTI)/tractography, prior to, immediately after, at one-month, 6-month, and 1-year follow-up status post-surgical resection. These data will also be collected at 18-month (±60 days) and 24-month (±60 days) visits post-surgery, if regular office visits with the neurosurgeon are scheduled at these two time points. Only at baseline, the following will be conducted: Brief Ataxia Rating Scale (BARS) assessment score, Cerebellar Cognitive Affective Scale (CCAS/Schmahmann syndrome) scale score, Montreal Cognitive Assessment (MoCA) assessment, and a quality of life (QoL) assessment using the SF-36 questionnaire.

Data analysis: For each test item within the CCAS there is a threshold score allowing a pass/fail determination that differentiates CCAS-positive patients from CCAS-negative patients. The primary, study endpoint is the percentage of patients with a positive CCAS diagnosis prior to surgery. The investigators will evaluate whether CCAS is preferentially seen in association with any demographic or descriptive variables (particularly tumor location in the cerebellum) using chi-squared testing unless otherwise indicated. Demographic data including sex, age at time of brain tumor diagnosis and at surgery, education level completed, and dominant writing hand will be described. The distribution of each of the following preoperative variables will also be described: presenting symptom (cognitive, motor, or vestibular), brain lesion type (newly diagnosed vs recurrent), primary tumor site, primary tumor histology, presence or absence of a systemic burden of disease, presence of hydrocephalus or previous seizure in 30 days prior to surgery, prior surgery, prior whole brain radiation or stereotactic radiosurgery, initiation of antiepileptic or steroids prior to surgery, the indication for surgery. These data will be used to compare baseline characteristic of cerebellar tumor patients with non-cerebellar brain tumor patients. All statistical analysis will be performed by the investigators using Prism 4.0 (GraphPad Software, Inc.) and Stata v10 (StataCorp Lp). Significance will be assessed at alpha = 0.05.

Risks/Benefits: There will be physical or health-related risks to the surgical resection of the patients' cerebellar tumor according to the standard of care. Risk is also involved to the extent that privacy and confidentiality may be compromised. However, every reasonable effort will be made to limit breaches of privacy and confidentiality. Participants will not benefit directly from this study. However, the results of this work will help improve the perioperative assessment of patients with tumors of the cerebellum, which may improve rehabilitation efforts in this unique patient population.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Patients with primary cerebellar brain tumors or metastatic brain tumors located in the cerebellum who will undergo surgery for tumor resection, OR with primary non-cerebellar brain tumors or metastatic tumors located in a non-cerebellar brain location who will undergo surgery for tumor resection

Exclusion Criteria:

* Patients under the age of 18
* Patients with intracranial pathologies (e.g. stroke, vasculitis, infection, developmental anomalies, etc.) outside of the cerebellum
* Non-oncologic cerebellar pathologies (e.g. stroke, vasculitis, infection, developmental anomalies, primary cerebellar ataxias, etc.)
* Patients who are illiterate, are blind, or do not read or understand English
* Patients with a Karnofsky Performance Status score of equal to less than 40

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Thirty-three adult (≥18 years of age) patients with primary cerebellar brain tumors or metastatic brain tumors located in the cerebellum who will undergo surgery for tumor resection, and 33 adult patients with primary non-cerebellar brain tumors or metastatic tumors located in a non-cerebellar brain location who will also undergo surgery for tumor resection will be included in this study. The non-cerebellar brain tumor control group will be included for comparison.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2021-02-28 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2027-05-17 (Estimated)

PRIMARY OUTCOMES:
Percentage of cerebellar tumor patients with a positive cerebellar cognitive affective syndrome (CCAS) diagnosis prior to surgery | Baseline
  CCAS/Schmahmann syndrome scale: 120 point scale (0=most severe cognitive impairment to 120=no cognitive impairment)
Percentage of brain non-cerebellar tumor patients with a positive cerebellar cognitive affective syndrome (CCAS) diagnosis prior to surgery | Baseline
  CCAS/Schmahmann syndrome scale: 120 point scale (0=most severe cognitive impairment to 120=no cognitive impairment)

SECONDARY OUTCOMES:
Neurological Impact of tumor location in patients undergoing resection of cerebellar tumors | Discharge (1-2 days after surgery)
  "Impact" will be determined with standard of care neurological evaluation and "tumor location" with magnetic resonance imaging (MRI) with or without diffusion tensor imaging (DTI)/tractography
Neurological Impact of tumor location in patients undergoing resection of cerebellar tumors | 1 month after surgery
  "Impact" will be determined with standard of care neurological evaluation and "tumor location" with magnetic resonance imaging (MRI) with or without diffusion tensor imaging (DTI)/tractography
Neurological Impact of tumor location in patients undergoing resection of cerebellar tumors | 6 months after surgery
  "Impact" will be determined with standard of care neurological evaluation and "tumor location" with magnetic resonance imaging (MRI) with or without diffusion tensor imaging (DTI)/tractography
Neurological Impact of tumor location in patients undergoing resection of cerebellar tumors | 12 months after surgery
  "Impact" will be determined with standard of care neurological evaluation and "tumor location" with magnetic resonance imaging (MRI) with or without diffusion tensor imaging (DTI)/tractography
Neurological Impact of tumor location in patients undergoing resection of cerebellar tumors | 18 months after surgery
  "Impact" will be determined with standard of care neurological evaluation and "tumor location" with magnetic resonance imaging (MRI) with or without diffusion tensor imaging (DTI)/tractography
Neurological Impact of tumor location in patients undergoing resection of cerebellar tumors | 24 months after surgery
  "Impact" will be determined with standard of care neurological evaluation and "tumor location" with magnetic resonance imaging (MRI) with or without diffusion tensor imaging (DTI)/tractography
Neurological Impact of tumor location in patients undergoing resection of brain non-cerebellar tumors | Discharge (1-2 days after surgery)
  "Impact" will be determined with standard of care neurological evaluation and "tumor location" with magnetic resonance imaging (MRI) with or without diffusion tensor imaging (DTI)/tractography
Neurological Impact of tumor location in patients undergoing resection of brain non-cerebellar tumors | 1 month after surgery
  "Impact" will be determined with standard of care neurological evaluation and "tumor location" with magnetic resonance imaging (MRI) with or without diffusion tensor imaging (DTI)/tractography
Neurological Impact of tumor location in patients undergoing resection of brain non-cerebellar tumors | 6 months after surgery
  "Impact" will be determined with standard of care neurological evaluation and "tumor location" with magnetic resonance imaging (MRI) with or without diffusion tensor imaging (DTI)/tractography
Neurological Impact of tumor location in patients undergoing resection of brain non-cerebellar tumors | 12 months after surgery
  "Impact" will be determined with standard of care neurological evaluation and "tumor location" with magnetic resonance imaging (MRI) with or without diffusion tensor imaging (DTI)/tractography
Neurological Impact of tumor location in patients undergoing resection of brain non-cerebellar tumors | 18 months after surgery
  "Impact" will be determined with standard of care neurological evaluation and "tumor location" with magnetic resonance imaging (MRI) with or without diffusion tensor imaging (DTI)/tractography
Neurological Impact of tumor location in patients undergoing resection of brain non-cerebellar tumors | 24 months after surgery
  "Impact" will be determined with standard of care neurological evaluation and "tumor location" with magnetic resonance imaging (MRI) with or without diffusion tensor imaging (DTI)/tractography

CONTACTS AND LOCATIONS:
Overall Officials: Allan H Friedman, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No